CLINICAL TRIAL: NCT06969248
Title: The Effects of Interventions Targeted to Fathers on Fathers' Participation in Infant Care, Attachment Status, and Paternal Depression: A Randomized Controlled Trial
Brief Title: Program to Increase Fathers' Involvement in Infant Care
Acronym: Infant Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Principal Investigator, Tuba Demirel, Assoc.Prof., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 9278; TUSEB (Other: Health Institutes of Türkiye)
Record Dates: First submitted 2025-03-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-03

CONDITIONS: Randomised Controlled Trial; Public Health Nursing; Child Health
Keywords: fathers' involvement in infant care; Edinburgh Postpartum Depression Scale.; Father-Infant Attachment; Child Health

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Since the trainings for the experimental group in the study will be conducted by the researcher conducting the study, researcher and participant blinding will not be possible. The data will be analyzed by an independent statistics expert. In this context, statistical blinding will be applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-Intervention Group (No Intervention): Fathers in the control group will continue their routine practices. Fathers in this group will be measured twice, pre-test and post-test. No intervention will be made to the control group. After the intervention group's training is completed, training contents and videos will be shared with the control group.
- Intervention Group (Experimental)
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — Fathers will be provided with a total of 8 weeks of training and videos. The training will cover the role of fatherhood and its historical development, the developmental stages and care needs of babies, ways for fathers to participate in baby care and the benefits of participation, father-infant bonding and influencing factors, and paternal depression. Videos on the subject will be shared with fathers.
  Arms: Intervention Group

SUMMARY:
Fathers participating in the study will be given an 8-week formality intervention. Participants will be shown 4-week infant care training records and then 4-week videos prepared on educational topics. The effect of the intervention will be determined annually by the mean scores of the Fathers' Participation in Infant Care Questionnaire, Father Infant Attachment Scale, and Edinburgh Postpartum Depression Scale.

DETAILED DESCRIPTION:
The study will be conducted in a Family Health Center in Turkey, selected by random lottery. Fathers who are registered in a family health center and have babies aged 4-12 months and fathers who have children for the first time will be included in the study. The type of the study is planned as randomized controlled pre-test post-test, parallel group experimental type. A total of 80 fathers will be included in the study, 40 in each group, according to the calculation made with Gpower analysis. Participants will be randomly assigned to groups. Nursing interventions will last for 8 weeks and participants will be given training and watched videos during this process.

ELIGIBILITY:
Inclusion Criteria

* Having a healthy baby between 4-12 months old,
* Being a first-time father,
* Volunteering to participate in the study,
* Having a smartphone

Exclusion Criteria:

* Being under 18 years old,
* Having a psychiatric diagnosis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Fathers' Involvement in Infant Care Questionnaire | 8 week
Father Infant Attachment Scale | 8 week
Edinburgh Postpartum Depression Scale | 8 week

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732